CLINICAL TRIAL: NCT03793114
Title: Residual Secretion of Adrenal Steroid Hormones in Addison's Disease
Brief Title: Screening and Stimulation Testing for Residual Secretion of Adrenal Steroid Hormones in Autoimmune Addison's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bergen (Other)
Collaborators: Karolinska Institutet (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2018/751/REK sør-øst A (REK)
Record Dates: First submitted 2018-11-06; First posted 2019-01-04 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Primary Adrenal Insufficiency
MeSH Terms: conditions — Addison Disease | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Detectable levels of adrenal hormones (Experimental): Patients with detectable serum levels of adrenal hormones will go through cosyntropin stimulation testing.
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- Controls with undetectable hormone levels (Active Comparator): Twenty patients without detectable serum levels of adrenal hormones will serve as controls in cosyntropin stimulation testing.
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- Undetectable levels of adrenal hormones (No Intervention): Patients without detectable serum levels of adrenal hormones. Cosyntropin stimulation testing will not be performed.
- Congenital adrenal hyperplasia (CAH) control group (Other): Mapping adrenal steroid profile in patients with congenital adrenal hyperplasia (CAH) with confirmed total deficiency of 21-hydroxylase.
  Interventions: Diagnostic Test: Baseline blood tests
- Bilaterally adrenalectomized control group (Other): Mapping adrenal steroid profile in patients who are bilaterally adrenalectomized.
  Interventions: Diagnostic Test: Baseline blood tests
- Diurnal variation in residual adrenocortical hormone levels (Experimental): Patients with detectable serum levels of adrenal hormones will go through a 30-hour ambulatory sampling of interstitial fluid for mapping of any diurnal variation in endogenous adrenocortical secretion.
  Interventions: Device: 30-hour ambulatory sampling of intestinal fluid
- Repeated cosyntropin testing in newly diagnosed patients (Experimental): Newly diagnosed patients will be invited to go through repeated cosyntropin testing to delineate the natural progression of adrenocortical failure.
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- Cardiovascular and inflammatory biomarkers (Active Comparator): Compare cardiovascular and inflammatory biomarker profiles in patients with and without residual production of adrenocortical steroids
  Interventions: Other: Blood test

INTERVENTIONS:
Diagnostic Test: Cosyntropin stimulation test — Blood samples are taken before (0 min), and 30 and 60 min after intravenously administration of 250 µg cosyntropin (tetracosactide acetate) with the patient placed in the recumbent position. The test will be performed non-fasting (but medication-fasting) between 08:00 and 10:00 a.m.
  Other Names: Synacthen stimulation test
  Arms: Controls with undetectable hormone levels; Detectable levels of adrenal hormones; Repeated cosyntropin testing in newly diagnosed patients
Diagnostic Test: Baseline blood tests — Medication-fasting morning levels of adrenocortical hormones.
  Arms: Bilaterally adrenalectomized control group; Congenital adrenal hyperplasia (CAH) control group
Device: 30-hour ambulatory sampling of intestinal fluid — 30-hour ambulatory sampling of intestinal fluid for analysis of adrenocortical hormones.
  Arms: Diurnal variation in residual adrenocortical hormone levels
Other: Blood test — Cardiovascular and inflammatory biomarker profiles
  Arms: Cardiovascular and inflammatory biomarkers

SUMMARY:
In autoimmune adrenal insufficiency, or Addison's disease (AD), the immune system attacks the adrenal cortex. As a result, the adrenal cells producing hormones such as cortisol and aldosterone are destroyed, leaving the body with insufficient levels to meet its needs. The common perception is that upon diagnosis of Addison's disease, basically all adrenal hormone production has ceased.

There have, however, been found a few individuals who preserve some residual secretion of cortisol even years after diagnosis. The objectives of this study is to find out how common it is, and to explore if residual function have impact on patient outcome. That is, do patients with and without residual function differ when it comes to quality of life, working ability, medication dosages, and risk of adrenal crisis?

DETAILED DESCRIPTION:
Autoimmune destruction of the adrenal cortex is the main cause of primary adrenal insufficiency (Addison's disease, AD). Autoimmune AD (AAD) becomes clinically manifest when 90 % of cortex of adrenal gland is destroyed. Current dogma says that adrenal insufficiency ultimately is complete, that is the adrenal cortex stops producing steroids altogether. However, several case reports indicate that there might be a subgroup of patients that retain some steroid production, even years after the diagnosis. This ability could be beneficial as it could protect against adrenal crises, ease medication, and leave the patient with better quality of life.

The objective of the study is to systematically assess to what extent patients with AAD have residual adrenocortical function, and to characterize this subgroup.

The study will be an open non-randomized three-stage multicenter clinical trial comprising patients from the Norwegian Registry for organ-specific autoimmune disease (ROAS), the Swedish Addison registry, and Germany. In stage 1, patients will be asked to fill out questionnaires and deliver medication-fasting samples for analyses of adrenal steroids. In addition, patients with congenital adrenal hyperplasia (CAH) and bilaterally adrenalectomized will serve as negative controls for adrenal steroids. In stage 2, AAD patients with residual steroid production will be invited to a cosyntropin stimulation test to estimate the maximum steroid output from the adrenal glands. Twenty patients with no sign of residual function will also be tested as a control group. In stage 3, AAD patients with confirmed residual function will be invited to go through a 30-hour ambulatory sampling of interstitial fluid for investigation of diurnal variation in adrenocortical hormone levels. Also, newly diagnosed AAD patients will be invited to repeated cosyntropin testing as a means of delineating the natural progression of adrenocortical failure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with AAD, age 18-70 years old. This requires documented adrenal insufficiency and a positive test for 21-hydroxylase autoantibodies (biomarker for autoimmune cause) on at least one occasion.
* Provided written informed consent
* In case of concomitant endocrine/autoimmune diseases, the patients should be on stable adequate treatment at least the last 3 months prior to the study period.
* For Norwegian AD patients: enrolled in ROAS
* For Swedish AD patients: enrolled in the Swedish Addison registry

Exclusion Criteria:

* Antihypertensive treatment, with the exception of doxazosin, verapamil, and moxonidine.
* Active malignant disease, severe heart, kidney or liver failure.
* Diabetes mellitus type 1.
* Pregnancy or breast feeding.
* Pharmacological treatment with glucocorticoids (except their usual cortisone or hydrocortisone replacement therapy) or drugs that interfere with cortisol and catecholamine metabolism (antiepileptics, rifampicin, St. Johns wart).
* Use of other glucocorticoid replacement medication than cortisone acetate or hydrocortisone.
* Intake of grapefruit, grapefruit juice, or and liquorice juice the last week before or during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of included patients with residual secretion of cortisol and aldosterone. | 1 day
  Percentage of included patients with detectable levels of adrenal steroid hormones.

SECONDARY OUTCOMES:
Medication-fasting adrenocorticotropic hormone (ACTH)-stimulated levels of metanephrines | 1 day
  Levels in blood samples
Medication-fasting basal levels of cortisol | 1 day
  Levels in blood samples
Medication-fasting basal levels of cortisol | 1 day
  Levels in urine samples
Medication-fasting basal levels of cortisol | 1 day
  Levels in hair samples
Medication-fasting basal levels of cortisol precursors | 1 day
  Levels in blood samples
Medication-fasting basal levels of cortisol precursors | 1 day
  Levels in urine samples
Medication-fasting basal levels of cortisol precursors | 1 day
  Levels in hair samples
Medication-fasting basal levels of cortisol metabolites | 1 day
  Levels in blood samples
Medication-fasting basal levels of cortisol metabolites | 1 day
  Levels in urine samples
Medication-fasting basal levels of cortisol metabolites | 1 day
  Levels in hair samples
Medication-fasting basal levels of aldosterone | 1 day
  Levels in blood samples
Medication-fasting basal levels of aldosterone | 1 day
  Levels in urine samples
Medication-fasting basal levels of aldosterone precursors | 1 day
  Levels in blood samples
Medication-fasting basal levels of aldosterone precursors | 1 day
  Levels in urine samples
Medication-fasting basal levels of aldosterone metabolites | 1 day
  Levels in blood samples
Medication-fasting basal levels of aldosterone metabolites | 1 day
  Levels in urine samples
Medication-fasting basal levels of renin in patients with and without residual function. | 1 day
  Levels in blood samples
Medication-fasting basal levels of renin in patients with and without residual function. | 1 day
  Levels in urine samples
Medication-fasting basal levels of ACTH in patients with and without residual function. | 1 day
  Levels in blood samples
Medication-fasting basal levels of ACTH in patients with and without residual function. | 1 day
  Levels in urine samples
Medication-fasting basal levels of metanephrines in patients with and without residual function | 1 day
  Levels in blood samples
Medication-fasting basal levels of metanephrines in patients with and without residual function | 1 day
  Levels in urine samples
Medication-fasting ACTH-stimulated levels of cortisol | 1 day
  Levels in blood samples
Medication-fasting ACTH-stimulated levels of cortisol precursors | 1 day
  Levels in blood samples
Medication-fasting ACTH-stimulated levels of cortisol metabolites | 1 day
  Levels in blood samples
Medication-fasting ACTH-stimulated levels of aldosterone | 1 day
  Levels in blood samples
Medication-fasting ACTH-stimulated levels of aldosterone precursors | 1 day
  Levels in blood samples
Medication-fasting ACTH-stimulated levels of aldosterone metabolites | 1 day
  Levels in blood samples
Cortisol replacement doses, including stress doses in patients with and without residual function. | 1 day
  Total daily dosage
Cortisol stress doses in patients with and without residual function. | 1 day
  No. stress doses the last week
Fludrocortisone replacement doses in patients with and without residual function. | 1 day
  Total daily dosage.
In patients with and without residual function: disease-specific quality-of-life | 1 day
  Total score ranging from 30 to 120 in disease-specific quality-of-life questionnaire, Addison Quality of Life (AddiQoL). For every question, scoring is translated in points (1 = 1 point, 2 and 3 = 2 points, 4 and 5 = 3 points, 6 = 4 points) and the algebraic sum of points is calculated. A higher score reflects better health-related quality-of-life.
In patients with and without residual function, generic health-related quality of life by the Short Form (36) Health Survey | 1 day
  The Short Form (36) Health Survey is a generic tool comprising 36 items evaluating patient reported quality of life concerning eight domains (physical functioning, role functioning physical, bodily pain, general health perception, vitality, social functioning, role functioning emotional, and mental health and general perception of change in health). Scores are expressed on a 0-100 scale with higher scores associated with better quality of life. The result of each domain is presented separately.
Number of adrenal crises pr. 100 patient years | 1 day
  Number of crises pr. 100 patient years for all included patients as well as in patients with versus without residual adrenal function

OTHER OUTCOMES:
Adrenocortical hormones in congenital adrenal hyperplasia (CAH) controls | 1 day
  Presence or absence of adrenocortical hormones in congenital adrenal hyperplasia (CAH) controls in a medication fasting morning baseline blood sample
Adrenocortical hormones in bilaterally adrenalectomized controls | 1 day
  Presence or absence of adrenocortical hormones in bilaterally adrenalectomized controls in a medication fasting morning baseline blood sample
Change in response to cosyntropin testing | 4 days
  Response to cosyntropin testing at 3, 6, 12, and 24 months after diagnosis
Diurnal variation in adrenocortical hormone secretion | 2 days
  Variation in endogenous adrenocortical hormone secretion during 30 hour continuous sampling

CONTACTS AND LOCATIONS:
Overall Officials: Eystein S Husebye, M.D, Prof, Principal Investigator — University of Bergen
Locations (3):
- Endokrinologie in Charlottenburg, Berlin, Germany
- Haukeland University Hospital, Bergen, Norway
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Upon informed and signed content, biological samples will be stored in the biobank for research on endocrine disorders. Any new analyses will not be performed without approval from the Regional committee for medical and health research ethics.

REFERENCES:
- [Derived] Saevik AB, Akerman AK, Methlie P, Quinkler M, Jorgensen AP, Hoybye C, Debowska AJ, Nedrebo BG, Dahle AL, Carlsen S, Tomkowicz A, Sollid ST, Nermoen I, Gronning K, Dahlqvist P, Grimnes G, Skov J, Finnes T, Valland SF, Wahlberg J, Holte SE, Simunkova K, Kampe O, Husebye ES, Bensing S, Oksnes M. Residual Corticosteroid Production in Autoimmune Addison Disease. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2430-41. doi: 10.1210/clinem/dgaa256. PMID 32392298